CLINICAL TRIAL: NCT06652191
Title: Effect of Central Venous Puncture Dilation and Non Dilation on the Success Rate of Catheterization
Brief Title: Non Dilation on the Central Venous Catheterization（NDCVC-01）
Acronym: NDCVC-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024ZSLYEC-387
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-07

CONDITIONS: the Success Rate of Non Dilation on the Central Venous Catheterization
Keywords: non-dilation; central venous catheterization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The test group:Direct catheterization with non-dilation (Experimental): Under the guidance of real-time ultrasound, the right internal jugular vein was punctured and a guide wire was inserted, place the catheter into the vessel directly along the guide wire without using an dilator to expand the skin
  Interventions: Procedure: Direct catheterization with non-dilation
- The control group: Catheterization after expanding the skin with a dilator (Active Comparator): Under the guidance of real-time ultrasound, the right internal jugular vein was punctured and a guide wire was inserted, after the skin is expanded with a dilator, the catheter is inserted into the vessel along the guide wire
  Interventions: Procedure: Catheterization after expanding the skin with a dilator

INTERVENTIONS:
Procedure: Direct catheterization with non-dilation — Under the guidance of real-time ultrasound, the right internal jugular vein was punctured and a guide wire was inserted, place the catheter into the vessel directly along the guide wire without using an dilator to expand the skin
  Arms: The test group:Direct catheterization with non-dilation
Procedure: Catheterization after expanding the skin with a dilator — Under the guidance of real-time ultrasound, the right internal jugular vein was punctured and a guide wire was inserted, after the skin is expanded with a dilator, the catheter is inserted into the vessel along the guide wire
  Arms: The control group: Catheterization after expanding the skin with a dilator

SUMMARY:
The central venous catheter is widely used and used in high dosage, and various complications such as hematoma, hemopneumothorax and arterial puncture may occur during puncture and use. In addition to conventional techniques, studies have been done to improve the success rate of puncture and reduce the incidence of complications by modifying different procedures. However, among the complications caused by the procedure of percutaneous catheter placement, the fatal bleeding caused by skin dilation may threaten the patient' s life. There are few studies on dilators and skin dilation steps at home and abroad. In this study, the conventional puncture technique was improved and the skin dilation step was omitted, hoping to reduce complications, reduce puncture time, improve efficiency and improve patient comfort on the premise of ensuring the success rate of catheterization.

DETAILED DESCRIPTION:
The Central venous catheter is widely used, but there are various complications. During the procedure of skin expansion with central venous catheterization, the use of a dilator can lead to complications such as hematoma, fatal bleeding, discomfort or serious threat to the patient's life. The aim of this study was to eliminate the procedure of skin expansion, to ensure the success rate of catheterization, to reduce complications, to reduce operation time, to improve efficiency, and to improve patients' comfort.

This study is a single-center, prospective, randomized controlled trial.The sample size was calculated by non-inferiority test:(1)the success rate of central venous catheterization was 97.98% according to Meta-analysis references;(2)α =0.025;(3)power 90%;(4)missed follow-up rate 20%, and ultimately 336 samples were included in the study,168 patients in each group.

Patients will receive written and verbal information about the trial before written consent is obtained. Randomization will take place on the day of surgery, and patients will be assigned to the intervention group (direct catheterization with non-dilation) or the control group (catheterization after expanding the skin with a dilator) . The randomization is performed using concealed allocation where envelopes are prepared externally using a randomization list prepared by a research assistant.

Under ultrasound guidance, The patient will undergo central venous catheterization by an experienced anesthesiologist based on grouping information.In the control group, catheter was inserted after skin expansion with dilator, while in the test group, catheter was inserted directly with non-dilator.The success rate of catheterization, the total time of catheterization, and complications were recorded.The patients were followed up for 24 hours after surgery and asked about their comfort level.

Shapiro-Wilk test is used to test normality for continuous variables, with data expressed as mean ± standard deviation, and independent t-test is used for statistical analysis.For categorical data, the incidence of immediate complications is expressed as a percentage (%), and chi square test is used to statistically analyze the incidence of various complications.For the Primary outcome ,success rate of catheterization, the method of confidence interval is used. If the lower limit of confidence interval > negative non-inferiority threshold, the non-inferiority is considered. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged 18 years or older
* (2) patients with internal jugular vein catheterization

Exclusion Criteria:

* （1）Patients with infection at the puncture site
* （2）Patients with contraindications to central venous catheterization
* （3）Patients with imaging examination suggesting thrombosis in the internal jugular vein before puncture
* （4）Patients who refused to participate, did not sign or refused to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Catheterization | Intraoperative (Start by locating the vessel until the catheter is confirmed to be in the target vessel)
  The ratio of the number of successful catheterization to the number of participants in each group.
  Confirm that the catheter in the target vessel is defined as:(1)The syringe smoothly draws back blood;(2)After the fluid is connected, the infusion drops flow smoothly

SECONDARY OUTCOMES:
Total time of catheterization | Intraoperative (Start with the tip of the needle touching the skin until the catheter is in the target) vessel
  This total time was defined as the time from the tip of the needle touching the skin to confirmation that the catheter was in the target vessel
Incidence of immediate complications | Intraoperative (Start by locating the vessel until the catheter is confirmed to be in the target vessel)
  immediate complications include：arterial puncture; pneumothorax; hemothorax; hematoma; Oozing blood; arrhythmia.
  definition: Arterial puncture : puncture of an artery with a needle during catheter placement.
  Pneumothorax :a collection of air or gas in the pleural cavity, which can cause the lung to collapse, confirmed by positive imaging.
  Hemothorax: a collection of blood in the pleural cavity, which can cause the lung to collapse, confirmed by positive imaging.
  hematoma: hematoma on the ultrasonography surrounding the vessel, severe hematoma defined as a visible hemotama large enough to be seen outside the skin.
  Oozing blood: Blood oozes from the skin at the point of puncture, or requiring dressing change.
  arrhythmia:a irregular heartbeat, include premature beats; atrial tachycardia; paroxysmal supraventricular tachycardia; atrial flutter; atrial fibrillation and so on.
Patient Comfort Score | 24 hours after catheterization
  Patients were assessed for comfort using the visual analogue scale(0-10). 0 was very uncomfortable, 10 was very comfortable, and the higher the score, the more comfortable the patient was.

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hostipal, Sun Yet Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] iData Research. Central Venous Catheter Market Size, Share & Trends Analysis, Global, 2020-2026. 2020. Accessed October 26, 2023
- [Result] 秦志均,等.改良中心静脉穿刺术对穿刺置管并发症的影响.现代临床医学2016( 04) :023
- [Result] Collier PE. Prevention and treatment of dilator injuries during central venous catheter placement. J Vasc Surg Venous Lymphat Disord. 2019 Nov;7(6):789-792. doi: 10.1016/j.jvsv.2019.06.020. Epub 2019 Aug 27. PMID 31471280
- [Result] Kulvatunyou N, Heard SO, Bankey PE. A subclavian artery injury, secondary to internal jugular vein cannulation, is a predictable right-sided phenomenon. Anesth Analg. 2002 Sep;95(3):564-6, table of contents. doi: 10.1097/00000539-200209000-00012. PMID 12198037
- [Result] Oropello JM, Leibowitz AB, Manasia A, Del Guidice R, Benjamin E. Dilator-associated complications of central vein catheter insertion: possible mechanisms of injury and suggestions for prevention. J Cardiothorac Vasc Anesth. 1996 Aug;10(5):634-7. doi: 10.1016/s1053-0770(96)80142-x. No abstract available. PMID 8841872
- [Result] Adhya S, Laha SK. Central venous catheterization. N Engl J Med. 2007 Aug 30;357(9):944; author reply 944-5. No abstract available. PMID 17806139
- [Result] Safety Committee of Japanese Society of Anesthesiologists. Practical guide for safe central venous catheterization and management 2017. J Anesth. 2020 Apr;34(2):167-186. doi: 10.1007/s00540-019-02702-9. Epub 2019 Nov 30. PMID 31786676
- [Result] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Result] Lim T, Ryu HG, Jung CW, Jeon Y, Bahk JH. Effect of the bevel direction of puncture needle on success rate and complications during internal jugular vein catheterization. Crit Care Med. 2012 Feb;40(2):491-4. doi: 10.1097/CCM.0b013e318232da48. PMID 21983370
- [Result] Lee YH, Kim TK, Jung YS, Cho YJ, Yoon S, Seo JH, Jeon Y, Bahk JH, Hong DM. Comparison of Needle Insertion and Guidewire Placement Techniques During Internal Jugular Vein Catheterization: The Thin-Wall Introducer Needle Technique Versus the Cannula-Over-Needle Technique. Crit Care Med. 2015 Oct;43(10):2112-6. doi: 10.1097/CCM.0000000000001167. PMID 26121076
- [Result] Kim E, Kim BG, Lim YJ, Jeon YT, Hwang JW, Kim HC, Choi YH, Park HP. A prospective randomised trial comparing insertion success rate and incidence of catheterisation-related complications for subclavian venous catheterisation using a thin-walled introducer needle or a catheter-over-needle technique. Anaesthesia. 2016 Sep;71(9):1030-6. doi: 10.1111/anae.13543. Epub 2016 Jul 11. PMID 27396474
- [Result] Song IK, Kim EH, Lee JH, Jang YE, Kim HS, Kim JT. Seldinger vs modified Seldinger techniques for ultrasound-guided central venous catheterisation in neonates: a randomised controlled trial. Br J Anaesth. 2018 Dec;121(6):1332-1337. doi: 10.1016/j.bja.2018.08.008. Epub 2018 Sep 7. PMID 30442261
- [Result] Teja B, Bosch NA, Diep C, Pereira TV, Mauricio P, Sklar MC, Sankar A, Wijeysundera HC, Saskin R, Walkey A, Wijeysundera DN, Wunsch H. Complication Rates of Central Venous Catheters: A Systematic Review and Meta-Analysis. JAMA Intern Med. 2024 May 1;184(5):474-482. doi: 10.1001/jamainternmed.2023.8232. PMID 38436976
- [Result] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Result] Smith RN, Nolan JP. Central venous catheters. BMJ. 2013 Nov 11;347:f6570. doi: 10.1136/bmj.f6570. No abstract available. PMID 24217269